CLINICAL TRIAL: NCT07284940
Title: Integrating Cognitive Elements Into Soccer Basic Skill Practice: Acute Effects on Cognitive Performance and Motor Learning
Brief Title: Cognitive-Integrated Soccer Training and Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fan Mao (Other)
Responsible Party: Sponsor-Investigator, Fan Mao, Clinical Professor, Qingdao University
Organization: Qingdao University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: QDU-HEC-2024376
Record Dates: First submitted 2025-11-20; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Executive Function (Cognition); Soccer Training; Performance; Motor Development
Keywords: integrative class; cognitive promotion; dribbling; soccer; physical education
MeSH Terms: conditions — Sialorrhea

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Only the coaches delivering the intervention are blinded to group allocation. Participants and outcome assessors are not blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitively Engaging Soccer Training (Experimental)
  Interventions: Behavioral: Cognitively Engaging Soccer Practice
- Conventional Soccer Training (Active Comparator)
  Interventions: Behavioral: Conventional Soccer Practice

INTERVENTIONS:
Behavioral: Cognitively Engaging Soccer Practice — This intervention integrates cognitive elements into basic soccer skill practice. Participants engage in 20-minute soccer dribbling sessions that include decision-making tasks, attention control, and working memory challenges embedded within motor actions. For example, players must react to color or number cues while performing dribbling drills. The purpose is to enhance both motor learning and cognitive performance through dual-task engagement.Cognitively Engaging Soccer Practice
  Arms: Cognitively Engaging Soccer Training
Behavioral: Conventional Soccer Practice — This intervention consists of traditional soccer dribbling training without added cognitive tasks. Participants perform the same duration and frequency of soccer skill practice (20 minutes) focusing purely on motor performance and technique refinement. No external cognitive demands are introduced.
  Arms: Conventional Soccer Training

SUMMARY:
This study aimed to examine the acute effects of integrating cognitive elements into basic soccer dribbling practice on cognitive performance and motor skill learning in adolescents.

A randomized controlled trial (RCT) was conducted involving 43 male adolescents, who were randomly assigned to either an experimental group or a control group. The experimental group participated in cognitively integrated dribbling practice, while the control group performed traditional cone-based dribbling practice. Each participant completed a single structured practice session lasting approximately 30 minutes.

Cognitive performance was assessed using the Flanker task and the 2-back task, while soccer skill learning was evaluated through standardized dribbling performance tests. All assessments were administered immediately before and after the practice session. The study was designed to compare short-term changes in cognitive and motor outcomes between the two training approaches under controlled conditions.

This trial contributes to understanding how cognitively enriched soccer practice may be structured and evaluated in adolescent populations within physical education and youth sport settings.

DETAILED DESCRIPTION:
The purpose of this study was to investigate whether incorporating cognitive elements into basic soccer dribbling drills influences cognitive task performance and motor skill learning in adolescents. Cognitive elements integrated into the practice were designed to engage processes such as attention control, inhibitory control, and working memory during motor execution.

The study employed a randomized controlled design with two parallel groups. Participants were randomly assigned to an experimental group, which performed cognitively integrated soccer dribbling drills, or a control group, which performed traditional soccer dribbling drills without explicit cognitive engagement. The intervention consisted of a single practice session lasting approximately 30 minutes.

Cognitive performance was evaluated using computerized versions of the Flanker task and the 2-back task. Motor skill learning was assessed using standardized soccer dribbling performance tests. All outcome measures were collected immediately before and after the intervention session to capture acute effects. The study design allows for controlled comparison of cognitive-integrated and traditional practice approaches in an adolescent population.

ELIGIBILITY:
Inclusion Criteria:

* Male adolescents aged 16-18 years;
* Healthy students with no recent injury affecting movement or physical activity;
* Normal or corrected-to-normal vision;
* Not taking any medication during the study period;
* Soccer novices with no formal or only limited soccer training experience

Exclusion Criteria:

* Diagnosed neurological disorders;
* Diagnosed musculoskeletal disorders;
* Use of medications known to affect cognitive function

Ages: 16 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Reaction time on cognitive tasks (Stroop task and 2-back task) | Baseline (pre-intervention, Day 1) and immediately post-intervention (Day 1)
  Reaction time (in milliseconds) will be recorded for correct responses during computerized Stroop and 2-back tasks. Mean reaction time across trials will be calculated separately for each task at each assessment time point.
Response accuracy on cognitive tasks (Stroop task and 2-back task) | Baseline (pre-intervention, Day 1) and immediately post-intervention (Day 1)
  Response accuracy will be calculated as the percentage of correct responses during computerized Stroop and 2-back tasks. Accuracy values will be summarized for each task at baseline and immediately after the intervention.

SECONDARY OUTCOMES:
Dribbling performance time | Baseline (pre-intervention, Day 1) and immediately post-intervention (Day 1)
  Dribbling performance time will be measured as the total time (in seconds) required to complete a standardized cone-dribbling course. The mean dribbling time will be calculated at baseline and immediately after the intervention to reflect short-term motor learning effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Qingdao University, School of Physical Education, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No
de-identified data available upon reasonable request

REFERENCES:
- [Result] Alesi M, Bianco A, Padulo J, Luppina G, Petrucci M, Paoli A, Palma A, Pepi A. Motor and cognitive growth following a Football Training Program. Front Psychol. 2015 Oct 27;6:1627. doi: 10.3389/fpsyg.2015.01627. eCollection 2015. PMID 26579014
- [Result] Mao F, Li Z, Qiu C, Fang Q. Developing integrative practice on basic soccer skills to stimulate cognitive promotion for children and adolescents. Front Psychol. 2024 Apr 19;15:1348006. doi: 10.3389/fpsyg.2024.1348006. eCollection 2024. No abstract available. PMID 38708011